CLINICAL TRIAL: NCT06198114
Title: Effects of Multi Sensory Integration on Hand Manipulation in Children With Visual Impairements
Brief Title: Effects of Multi Sensory Integration on Visual Impaired Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0746
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Visual Impairment
Keywords: Visual Impairment; Multi Sensory Integration
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi Sensory Integration (Experimental): This group will be treated with activity based training In which place different( nuts, screws, bullets, coins, paper clips, coloring ,scissor cutting with different shapes , Simulated feeding (by collecting beans with a spoon and transferring them into a container),transfer light and heavy weight objects into empty box.
  Interventions: Other: Multi Sensory Therapy
- Conventional Therapy (Active Comparator): This group will be treated with traditional therapy in which Place toys/objects inside and encourage the student to reach in and pull them out as well as put them back in. Give the student objects that can be put together and pulled apart. Encourage the students to use two hands in an organized manner to manipulate objects (e.g., grasp/release, twist/turn, rotate and examine, open/close, stack, nest).
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Multi Sensory Therapy — This group will be treated with activity based training by place different( nuts, screws, bullets, coins, paper clips, coloring ,scissor cutting with different shapes , Simulated feeding (by collecting beans with a spoon and transferring them into a container),transfer light and heavy weight objects into empty box. 5 days in a week
  Arms: Multi Sensory Integration
Other: Conventional Therapy — This group will be treated with traditional therapy in which Place toys/objects inside and encourage the student to reach in and pull them out as well as put them back in. Give the student objects that can be put together and pulled apart. Encourage the students to use two hands in an organized manner to manipulate objects (e.g., grasp/release, twist/turn, rotate and examine, open/close, stack, nest).5 days a week for an hour/daily.
  Arms: Conventional Therapy

SUMMARY:
Visual impairment is use to describe any kind of vision loss, whether it's someone who cannot see at all or someone who has partial vision loss. visual impairment is classified on the bases of visual acuity like mild, moderate, severe, profound, near total visual impairment, no light perception (NLP). Multisensory integration refers to a broad class of computations involving multiple sensory modalities in which information is integrated to produce an enhanced (or degraded) response.A Randomized control trail will be conducted at rising sun institute for disable children. Total sample size will be of 40 participants. After meeting the inclusion and exclusion criteria participants will be divided into two groups .Group A Control group will receive conventional therapy program. Place toys/objects inside and encourage the student to reach in and pull them out as well as put them back in. Give the student objects that can be put together and pulled apart. Group B will be treated with standard activity based therapy In which place different( nuts, screws, bullets, coins, paper clips, coloring ,scissor cutting with different shapes, Simulated feeding (by collecting beans with a spoon and transferring them into a container),transfer light and heavy weight objects into empty box. Nine whole peg tests are used to measure fine dexterity in visual impaired children. Jebsen Taylor hand function test for quantify motor hand function test. Total time for treatment per session will 45 minutes and duration of treatment will be 12 weeks, four days a week.box and block test used to improve manual hand dexterity. Assessment will be taken pre treatment, mid treatment at 4th week and 8th week and post treatment after 12th week. Data will be analyzed by SPSS

DETAILED DESCRIPTION:
Group(A)Will be treated with traditional therapy in which Place toys/objects inside and encourage the student to reach in and pull them out as well as put them back in. Give the student objects that can be put together and pulled apart. Encourage the students to use two hands in an organized manner to manipulate objects (e.g., grasp/release, twist/turn, rotate and examine, open/close, stack, nest).5 days a week for an hour/daily .Group(B)Will be treated with activity based training by place different( nuts, screws, bullets, coins, paper clips, coloring ,scissor cutting with different shapes , Simulated feeding (by collecting beans with a spoon and transferring them into a container),transfer light and heavy weight objects into empty box. 5 days in a week.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female age from( 05 -12year)
* Children from a Special Education School
* Visual acuity is 20/200 and check by hytos visual function test(9).
* All participants are label with legally blind by an ophthalmologist.
* Experienced physician screened the all participants and gave the good remark for the participation in training program.

Exclusion Criteria:

* Other History of neurological or developmental disorders
* Medical conditions that may affect motor development
* Inability to follow instructions or participate in study tasks
* Incomplete data or missing information
* Factors that could affect the validity or generalizability of the study findings Illness or Infection.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
BOX AND BLOCK TEST | 8 weeks
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations, including clients with visual impairment. The BBT is composed of a wooden box divided in two compartments by a partition and 150 blocks. The BBT administration consists of asking the client to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds. Higher score of transferring block into another box in 60 second determined the hand dexterity
HOYT'S FUNCTION TEST | 8 weeks
  Hoyt's level of visual function used to determine visual functional level before starting treatment.
JEBSEN TAYLOR HAND FUNCTION TEST: | 8 weeks
  The test includes tasks that assess fine hand motor function and functional tasks with and without weight. It consists of seven subtests, which are performed on time. We used different (nuts, bullets, heavy and light objects , different metals bottle cap) The score for the subtest is equal to the time in seconds required to complete the task, the maximum score for the subtest is 120. The total score is equal to the sum of points for all subtests and is calculated separately for each hand. The Higher the score, the better the child's hand function. Time will be 40 minutes with 2 Session Per week over the periods of 08 weeks
NINE HOLE PEG TEST | 8 weeks
  The test includes task that asses fine hand motor function and functional tasks. In which we use different objects like Board (wood or plastic), container for the pegs ,9 pegs, stopwatch .Instruct the patient to take the pegs from a container, one by one, and place them into the holes on the board, as quickly as possible, using only the hand being evaluated. Then, instruct the patient to remove the pegs from the holes, one by one, and replace them back into the container. The evaluator should start the stopwatch as soon as the patient touches the first peg. The evaluator should stop the stopwatch once the last peg is in the container. The number of seconds it takes for the patient to complete the test. Alternative scoring - the number of pegs placed in 50 or 100 seconds can be recorded. In this case, results are expressed as the number of pegs placed per second

CONTACTS AND LOCATIONS:
Overall Officials: Maria Munawar, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cemali M, Pekcetin S, Aki E. The Effectiveness of Sensory Integration Interventions on Motor and Sensory Functions in Infants with Cortical Vision Impairment and Cerebral Palsy: A Single Blind Randomized Controlled Trial. Children (Basel). 2022 Jul 27;9(8):1123. doi: 10.3390/children9081123. PMID 36010014
- [Background] Gori M. Multisensory Integration and Calibration in Children and Adults with and without Sensory and Motor Disabilities. Multisens Res. 2015;28(1-2):71-99. doi: 10.1163/22134808-00002478. PMID 26152053